CLINICAL TRIAL: NCT04270773
Title: Immunogenicity and Safety of a 9-valent Human Papillomavirus Vaccine in HIV-positive Women.
Acronym: 9-VPH-MVIH
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Virgen de las Nieves (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Carmen Hidalgo Tenorio, Principal Investigator, University Hospital Virgen de las Nieves
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9-VPH-MVIH
Record Dates: First submitted 2020-01-13; First posted 2020-02-17 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: HIV Infections; HPV Infection
MeSH Terms: conditions — HIV Infections; Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Intervention Model Description: This is a phase IV (post-authorization study), open, single-arm trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Only arm (Other): Single arm, Receiving treatment
  Interventions: Biological: Human Papillomavirus 9-valent Vaccine, Recombinant

INTERVENTIONS:
Biological: Human Papillomavirus 9-valent Vaccine, Recombinant — Vaccine administrated

SUMMARY:
In adult HIV-positive patients, data on the safety and immunogenicity of the quadrivalent HPV (qHPV) vaccine have been reported with excellent results (13 14); also, the results of a clinical trial of qHPV vaccine conducted in seropositive patients older than 36 years (WLHIV and MSM) have been published.

Even now, there is not a trial about immunogenicity and safety of a 9-valent human papillomavirus vaccine in HIV-positive women; for this reason, the investigators plan to conduct this clinical trial.

HYPOTHESYS: The administration of Nonavalent HPV vaccine (HPV-9) in adult women living with HIV will produce antibodies against nine genotypes of HPV, thus preventing the acquisition of new infections by those genotypes. Besides, this will prevent the cervical and anal dysplasia in these women.

DETAILED DESCRIPTION:
This is a phase IV (post-authorization study), open, single-arm trial of 9-valent human papillomavirus (9-HPV) vaccine in HIV-positive women. The recruitment and follow-up period will be 6 and 30 months, respectively.

At the initial clinical visit (V0), the conditions and objectives of the study were explained. The details were summarised in a document, which was presented to the patient who then signed the informed consent form. 2 mucosa samples were taken from the anal canal for the detection and genotyping of the HPV and for anal cytology; and high resolution anoscopy will be carried out. The patients will send to gynaecologist for exploration. Finally, full blood haemogram and blood chemistry analysis were measured, together with cluster of differentiation 4 (CD4), cluster of differentiation 8 (CD8) lymphocytes counts, HIV viral load (VL) and antibodies against 9 genotypes of the 9-HPV vaccine. 9-HPV vaccine will be administered at day 1 (V1), month 2 (V2) and month 6 (V3). Flow of subjects through the study in graphic 1.

Settings and locations: The patients who enrolled were HIV-positive women that were attending the Infectious Diseases Service of the "University Hospital Virgen de las Nieves", Granada (Spain), "Hospitalary Complex Ciudad de Jaén" (Spain) and "University hospital San Cecilio", Granada (Spain).

The purposes of the study were explained to the potential participants who then underwent screening, and enrolled if they met the inclusion criteria for the trial. They were asked to sign the fully informed consent form. The study will be conducted in compliance with ethical and moral principles stated in the Declaration of Helsinki as well as the current Spanish Laws on Biomedical Research(LEY 14/2007, de 3 de julio). Data were coded to ensure anonymity.

SAMPLE SIZE CONSIDERATIONS:

Currently, the rate of infections in unvaccinated women in the participating centers is 46.4% (12). The efficacy rate of the tetravalent vaccine in the prevention of cervical cancer is close to 100% and in the appearance of external anal lesions in men, around 85% (21). Considering that in our study population, the effectiveness is at least 75%, to achieve an accuracy of 5% in the estimation of a proportion through a normal 95% asymptotic confidence interval, assuming that the proportion is 11, 6% (25% of 46.4%), it will be necessary to include 158 women in the study. To this sample size will be added 10% in anticipation of possible losses in the follow-up or dropouts.

DATA COLLECTION:

All data were collected and coded to ensure anonymity according to the current legal requirements in Spain and European Union (EU) (GDPR Regulation (EU) 2016/679). At the initial clinical visit (V0), the conditions and objectives of the study were explained to subjects. The details were summarised in a document, which was presented to the patient who then signed the informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive women patients of ≥18 years of age who, at the time of study inclusion were not infected simultaneously by the 16, 18 genotypes of HPV in vagina and/or anus.

Exclusion Criteria:

* WLHIV patients who had simultaneous anal infection with the 16, 18, 31, 33, 45, 52 y 58 genotypes. - WLHIV diagnosed in V0 of ASCC or anal HSIL.
* Active opportunist infection at the time of recruitment into the study.
* Cd4 count < 200 cel/µL.
* History of allergy to aluminium and/or yeast extract excipient.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Antibodies against the 9 genotypes of the qHPV vaccine | 30 months
  immunogenicity of a 9-valent human papillomavirus vaccine in HIV-positive women older than ≥18 years
Incidence of Treatment-Emergent Adverse Events of a 9-valent human papillomavirus vaccine in HIV-positive women older than ≥18 years | Through study completion, up to 30 months
  Number of Participants With Any Adverse Event (AE)

SECONDARY OUTCOMES:
new HPV genotypes | Determined at 12th, 24th, 30th month
  acquisition rate of HPV genotypes of anal and cervical mucosa.
Data analysis of risk factors in subject who acquire HPV genotypes from data recorded at follow-up visits via survey. | 30 months
  The survey asks about HPV risk factors.
progression to dysplastic lesions | Determined at 12th, 24th, 30th month
  rate of progression to dysplastic lesions (LSIL, high grade squamous intraepithelial lesion (HSIL) and Cancer) anal and cervical after vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen de Las Nieves, Granada, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Palefsky JM. Human papillomavirus-associated anal and cervical cancers in HIV-infected individuals: incidence and prevention in the antiretroviral therapy era. Curr Opin HIV AIDS. 2017 Jan;12(1):26-30. doi: 10.1097/COH.0000000000000336. PMID 27828801
- [Background] Stier EA, Sebring MC, Mendez AE, Ba FS, Trimble DD, Chiao EY. Prevalence of anal human papillomavirus infection and anal HPV-related disorders in women: a systematic review. Am J Obstet Gynecol. 2015 Sep;213(3):278-309. doi: 10.1016/j.ajog.2015.03.034. Epub 2015 Mar 19. PMID 25797230
- [Background] Jemal A, Simard EP, Dorell C, Noone AM, Markowitz LE, Kohler B, Eheman C, Saraiya M, Bandi P, Saslow D, Cronin KA, Watson M, Schiffman M, Henley SJ, Schymura MJ, Anderson RN, Yankey D, Edwards BK. Annual Report to the Nation on the Status of Cancer, 1975-2009, featuring the burden and trends in human papillomavirus(HPV)-associated cancers and HPV vaccination coverage levels. J Natl Cancer Inst. 2013 Feb 6;105(3):175-201. doi: 10.1093/jnci/djs491. Epub 2013 Jan 7. PMID 23297039
- [Background] Firnhaber C, Westreich D, Schulze D, Williams S, Siminya M, Michelow P, Levin S, Faesen M, Smith JS. Highly active antiretroviral therapy and cervical dysplasia in HIV-positive women in South Africa. J Int AIDS Soc. 2012 Jun 7;15(2):17382. doi: 10.7448/IAS.15.2.17382. PMID 22713259
- [Background] Piketty C, Selinger-Leneman H, Grabar S, Duvivier C, Bonmarchand M, Abramowitz L, Costagliola D, Mary-Krause M; FHDH-ANRS CO 4. Marked increase in the incidence of invasive anal cancer among HIV-infected patients despite treatment with combination antiretroviral therapy. AIDS. 2008 Jun 19;22(10):1203-11. doi: 10.1097/QAD.0b013e3283023f78. PMID 18525266
- [Background] Franceschi S, Lise M, Clifford GM, Rickenbach M, Levi F, Maspoli M, Bouchardy C, Dehler S, Jundt G, Ess S, Bordoni A, Konzelmann I, Frick H, Dal Maso L, Elzi L, Furrer H, Calmy A, Cavassini M, Ledergerber B, Keiser O; Swiss HIV Cohort Study. Changing patterns of cancer incidence in the early- and late-HAART periods: the Swiss HIV Cohort Study. Br J Cancer. 2010 Jul 27;103(3):416-22. doi: 10.1038/sj.bjc.6605756. Epub 2010 Jun 29. PMID 20588274
- [Background] Hidalgo-Tenorio C, de Jesus SE, Esquivias J, Pasquau J. High prevalence and incidence of HPV-related anal cancer precursor lesions in HIV-positive women in the late HAART era. Enferm Infecc Microbiol Clin (Engl Ed). 2018 Nov;36(9):555-562. doi: 10.1016/j.eimc.2017.10.014. Epub 2017 Dec 6. English, Spanish. PMID 29208455
- [Background] Hidalgo-Tenorio C, Rivero-Rodriguez M, Gil-Anguita C, Esquivias J, Lopez-Castro R, Ramirez-Taboada J, de Hierro ML, Lopez-Ruiz MA, Martinez RJ, Llano JP. The role of polymerase chain reaction of high-risk human papilloma virus in the screening of high-grade squamous intraepithelial lesions in the anal mucosa of human immunodeficiency virus-positive males having sex with males. PLoS One. 2015 Apr 7;10(4):e0123590. doi: 10.1371/journal.pone.0123590. eCollection 2015. PMID 25849412
- [Background] Park IU, Palefsky JM. Evaluation and Management of Anal Intraepithelial Neoplasia in HIV-Negative and HIV-Positive Men Who Have Sex with Men. Curr Infect Dis Rep. 2010 Mar;12(2):126-33. doi: 10.1007/s11908-010-0090-7. Epub 2010 Feb 24. PMID 20461117
- [Background] Wilkin T, Lee JY, Lensing SY, Stier EA, Goldstone SE, Berry JM, Jay N, Aboulafia D, Cohn DL, Einstein MH, Saah A, Mitsuyasu RT, Palefsky JM. Safety and immunogenicity of the quadrivalent human papillomavirus vaccine in HIV-1-infected men. J Infect Dis. 2010 Oct 15;202(8):1246-53. doi: 10.1086/656320. PMID 20812850
- [Background] Wilkin TJ, Chen H, Cespedes MS, Leon-Cruz JT, Godfrey C, Chiao EY, Bastow B, Webster-Cyriaque J, Feng Q, Dragavon J, Coombs RW, Presti RM, Saah A, Cranston RD. A Randomized, Placebo-Controlled Trial of the Quadrivalent Human Papillomavirus Vaccine in Human Immunodeficiency Virus-Infected Adults Aged 27 Years or Older: AIDS Clinical Trials Group Protocol A5298. Clin Infect Dis. 2018 Oct 15;67(9):1339-1346. doi: 10.1093/cid/ciy274. PMID 29659751
- [Background] Hidalgo-Tenorio C, Ramirez-Taboada J, Gil-Anguita C, Esquivias J, Omar-Mohamed-Balgahata M, SamPedro A, Lopez-Ruz M, Pasquau J. Safety and immunogenicity of the quadrivalent human papillomavirus (qHPV) vaccine in HIV-positive Spanish men who have sex with men (MSM). AIDS Res Ther. 2017 Jul 18;14(1):34. doi: 10.1186/s12981-017-0160-0. PMID 28720147